CLINICAL TRIAL: NCT06989164
Title: Quantifying Differential Individual Responses to OGTT, Starchy Foods, and Mitigators and Its Association With Metabolic Subphenotypes
Brief Title: Post Prandial Individual Responses to Different Foods
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Yue Wu, Post doctoral, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 80689
Record Dates: First submitted 2025-05-13; First posted 2025-05-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: PreDiabetes; Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Participants will be asked to consume pre-portioned foods on different days as the first meal of the day, use a CGM, and take saliva and micro samples of blood before and after each meal. Food, supplements, and short exercise will be tested to see the post prandial effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diet Cycles (Experimental): Participants will be asked to consume pre-portioned foods on different days as the first meal of the day, use a CGM, and take saliva and micro samples of blood before and after each meal.
  Interventions: Other: Post prandial testing

INTERVENTIONS:
Other: Post prandial testing — A variety of foods, supplements, and short prescriptive exercise will be tested to see which one helps mitigate the rise is postprandial glucose after eating carbohydrate containing foods.

SUMMARY:
This study aims to understand why people respond differently to the same foods, especially when it comes to changes in blood sugar after eating. A continuous glucose monitors (CGMs) will be used to observe how individuals respond to specific meals and drinks (e.g., Oral Glucose Tolerance Test, OGTT). By studying these patterns, the investigators hope to identify different types of metabolism and see if certain foods or food ingredients (like fiber, amino acids, or vinegar) can help control blood sugar better for specific groups. This research will help lay the groundwork for personalized dietary advice based on a person's unique biology.

DETAILED DESCRIPTION:
Participants in the study will be provided with a continuous glucose monitor (CGM) and pre-measured cooked rice to test with different potential mitigators: fiber, acid, amino acid (e.g., leucine), whole protein, and exercise. Each of these conditions will be tested on a different day following strict instructions. For some of these tests, participants will be asked to collect a blood microsample and a saliva sample before and after eating the test meal. A stool sample will be collected at baseline.

ELIGIBILITY:
Inclusion Criteria:

* BMI (body mass index) >19 kg/m2 but < 45 kg/m2
* HbA1c < or equal to 7.0% while not on antihyperglycemic medications
* Be willing to provide written informed consent for all study procedures.
* Able to commute to Stanford campus for on-site visits

Exclusion Criteria:

* recent (<6mos) CVD (cardiovascular disease) event
* active malignancy
* kidney/liver disease
* pregnancy/lactation
* chronic inflammatory disease
* eating disorder
* bariatric surgery
* history of acute pancreatitis
* current use of antihyperglycemic, diabetogenic, or weight loss medications
* heavy alcohol use
* physical activity >2 hours/day
* inability to come to Stanford CTRU (Clinical and Translational Research Unit) for metabolic testing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Post prandial peak glucose levels | 3 hours
  Delta glucose peak within 3 hours after consuming the standard meal - peak glucose value minus baseline glucose value at time 0 measured by CGM in mg/dL.
Post prandial glucose area under the curve (AUC) | 3 hours
  AUC (>baseline) within three hours measured by CGM in mg/dL during the 3 hours after each study meal.

SECONDARY OUTCOMES:
Glucose time to peak | 3 hours
  The time in minutes from baseline to peak within 3 hours measured by CGM after each standardized meal.
Changes in personal post prandial metabolic states as measured in micro-sampling by targeted and untargeted metabolomics (LC-MS) | 1 hour
  Dry blood samples will be collected by micro-sampling before and 1 hour after the standardized meals. Based on those samples, metabolomics (e.g., short-chain fatty acids, amino acids and other polar and nonpolar metabolites) will be extracted and quantified by liquid chromatography mass spectrometry (LC-MS). Both hydrophilic LC and reverse phase LC will be used. Q Exactive will be used for MS. Tandem MS will be collected for annotation. Relative quantification will be used, where the level of metabolites can be compared between samples. Chemical reference will be used for the absolute quantification of targeted metabolites.
Individual microbiome composition | Baseline
  Microbiome will be defined by using metagenomics assay to baseline samples
Changes in postprandial proteomic responses as measured in micro-sampling by Olink | 1 hour
  Dry blood samples will be collected by micro-sampling frequently before and after the standardized meals. Based on those samples, proteomics will be quantified by proximity extension assay for the cardiometabolic panel. 96 proteins will be measured in the unit of normalized protein expression.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigator plan to share de-identified data to both public repositories and integrated databases when the consent of data sharing is obtained. The analysis results will be shared with the publication.
Time Frame: De-identified data will be shared with the future publications.
Access Criteria: De-identified data will be shared in public repositories. Metabolomics, microbiome, proteomics, and CGM measured glycemic response will be open to public access through the corresponding repositories.